CLINICAL TRIAL: NCT01761916
Title: Randomized Clinical Trial for Effectiveness of Clonidine Versus Captopril for Treatment of Postpartum Very High Blood Pressure
Brief Title: Clonidine Versus Captopril for Treatment of Postpartum Very High Blood Pressure
Acronym: CLONCAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Materno Infantil Prof. Fernando Figueira (Other)
Responsible Party: Principal Investigator, Leila Katz, MD pHD, Instituto Materno Infantil Prof. Fernando Figueira
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLONCAP
Record Dates: First submitted 2012-10-30; First posted 2013-01-07 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-06

CONDITIONS: Preeclampsia
Keywords: captopril, clonidine, pregnancy-induced hypertension,
MeSH Terms: conditions — Pre-Eclampsia; Hypertension, Pregnancy-Induced | interventions — Clonidine; Captopril

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CLONIDINE (Experimental): Postpartum patients with very high blood pressure will be treated with oral clonidine (0,1mg)
  Interventions: Drug: CLONIDINE
- CAPTOPRIL (Active Comparator): Postpartum patients with very high blood pressure will be treated with oral CAPTOPRIL (25mg)
  Interventions: Drug: CAPTOPRIL

INTERVENTIONS:
Drug: CLONIDINE — Postpartum patients with very high blood pressure will be treated with oral clonidine (0,1mg)
  Other Names: CLON
  Arms: CLONIDINE
Drug: CAPTOPRIL — Postpartum patients with very high blood pressure will be treated with oral captopril (25mg)
  Other Names: CAP
  Arms: CAPTOPRIL

SUMMARY:
The postpartum period represents a stage of the pregnancy-puerperal still rarely addressed scientifically. There are no reports in the literature and concrete enough to elucidate important issues, especially in the field of hypertension and pregnancy.

Searches based on current evidence concentrate their focus on the diagnosis of hypertensive disorders and treatment of these diseases maternofetais repercussions. However, the prognosis in the short and long term, as the BP outcome in mothers with severe preeclampsia, the most effective treatment for the control of hypertensive crisis and metabolic and cardiovascular events after two years of termination of pregnancy require further clarification.

The main idea for developing this research came from the clinical experience with the use of captopril in Obstetric ICU IMIP. This drug has long been used in postpartum women with severe preeclampsia or chronic hypertension exacerbated by pregnancy for control of hypertensive crisis and keeping pressure levels. Following the technical standards of the institution and during his administration, there were reports of side effects such as dry cough and nausea, beyond the threshold dose of 150mg daily captopril was easily achieved hindering control the use of hypotensive.

Alternative therapy, clonidine began to be used in mothers with some restriction on the use of ACE inhibitors and its hypotensive effect for peak pressure was satisfactory. What is not known yet is how long clonidine reduces high blood pressure and how long to leave stabilized compared to the use of captopril.

There are no reports in the literature databases, no randomized clinical trials that prove the effectiveness of clonidine for the treatment of hypotensive pressure peaks in this particular group of patients, even in comparison with other classes of antihypertensive drugs, especially captopril, to this purpose.

The investigators' primary assumption is that clonidine has better effectiveness in decreasing the frequency of pressure peaks when compared with captopril.

DETAILED DESCRIPTION:
The postpartum period represents a stage of the pregnancy-puerperal still rarely addressed scientifically. There are no reports in the literature and concrete enough to elucidate important issues, especially in the field of hypertension and pregnancy.

Searches based on current evidence concentrate their focus on the diagnosis of hypertensive disorders and treatment of these diseases maternofetais repercussions. However, the prognosis in the short and long term, as the BP outcome in mothers with severe preeclampsia, the most effective treatment for the control of hypertensive crisis and metabolic and cardiovascular events after two years of termination of pregnancy require further clarification.

The main idea for developing this research came from the clinical experience with the use of captopril in Obstetric ICU IMIP. This drug has long been used in postpartum women with severe preeclampsia or chronic hypertension exacerbated by pregnancy for control of hypertensive crisis and keeping pressure levels. Following the technical standards of the institution and during his administration, there were reports of side effects such as dry cough and nausea, beyond the threshold dose of 150mg daily captopril was easily achieved hindering control the use of hypotensive.

Alternative therapy, clonidine began to be used in mothers with some restriction on the use of ACE inhibitors and its hypotensive effect for peak pressure was satisfactory. What is not known yet is how long clonidine reduces high blood pressure and how long to leave stabilized compared to the use of captopril.

There are no reports in the literature databases, no randomized clinical trials that prove the effectiveness of clonidine for the treatment of hypotensive pressure peaks in this particular group of patients, even in comparison with other classes of antihypertensive drugs, especially captopril, to this purpose.

The investigators' primary assumption is that clonidine has better effectiveness in decreasing the frequency of pressure peaks when compared with captopril.

A triple blind randomized clinical trial will be conducted. Postpartum women with hypertensive disorders of pregnancy, admitted to the obstetric ICU of IMIP will be included in the research. After inclusion in the study, drugs for for very high blood pressure, according to randomization(captopril and clonidine)will be used. clonidine and captopril are administered at a dose of 25mg and 0.1mg respectively. If there is no control of blood pressure in 20 minutes new hypotensive doses will be administered until a total of 150mg/day (six tablets) and Captopril 0.6 mg / day (six tablets) clonidine. After exceeded the allowed dose, other drugs may be associated. Initially, nifedipine (30mg/day to 60mg/day) according to the service routine. The goal of intervention is to maintain a systolic blood pressure below 170mmHg and diastolic pressure below 110mmHg, with the lowest possible dose. Thus, these medications will be increased should the need arise, according to measurements taken daily by the attending physician and the nursing staff.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive disorders of pregnancy;
* Postpartum;
* Age 18 to 45 years;
* Very high blood pressure

Exclusion Criteria:

* Cardiac disease;
* Smoking;
* Use of illicit drugs that may interfere with maternal hemodynamics;
* Contraindications to the use of captopril: renal failure, chronic liver disease and hypersensitivity to the drug;
* Contraindications to the use of clonidine: sinus node disease, chronic liver disease and hypersensitivity to the drug;
* Inability to receive postpartum oral medications

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Time until resolution of very high blood pressure episode | During hospital stay, up until one month postpartum
  The time until resolution of very high blood pressure episode after clonidin or captopril use.

SECONDARY OUTCOMES:
Maternal outcomes | During hospital stay, up until one month postpartum
  Daily average systolic blood pressure;Daily average diastolic blood pressure;Need for combination with other hypotensive agent for the peak pressure or antihypertensive treatment maintenance;Need for new dose of antihypertensive medication for very high blood pressure; Laboratory tests during the postpartum; Adverse effects of hypotensive used for very high blood pressure;Puerperal complications

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Noronha, MD, Principal Investigator — IMIP
Locations (1):
- IMIP, Recife, Pernambuco, Brazil

REFERENCES:
- [Derived] Noronha Neto C C, Maia SS, Katz L, Coutinho IC, Souza AR, Amorim MM. Clonidine versus Captopril for Severe Postpartum Hypertension: A Randomized Controlled Trial. PLoS One. 2017 Jan 26;12(1):e0168124. doi: 10.1371/journal.pone.0168124. eCollection 2017. PMID 28125624
- [Derived] Noronha-Neto C, Katz L, Coutinho IC, Maia SB, Souza AS, Amorim MM. Clonidine versus captopril for treatment of postpartum very high blood pressure: study protocol for a randomized controlled trial (CLONCAP). Reprod Health. 2013 Jul 30;10:37. doi: 10.1186/1742-4755-10-37. PMID 23899372